CLINICAL TRIAL: NCT01541267
Title: The Effect of Various Types of the Renin-angiotensin-aldosterone System Blockade on Proteinuria in Chronic Non-diabetic Kidney Disease: a Double-blind Cross-over Randomised Controlled Study
Brief Title: The Effect of Various Types of the Renin-angiotensin-aldosterone System Blockade on Proteinuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Leszek Tylicki, MD PhD, Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ST-4/Aliskiren/2011
Record Dates: First submitted 2012-02-11; First posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: aliskiren; eplerenon; telmisartan; direct renin inhibitor; ACE inhibitor; mineralocorticoid inhibitor; proteinuria; chronic kidney diseases; renin-angiotensin-aldosterone system
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — aliskiren; Eplerenone; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C - A - B (Active Comparator): (A) telmisartan 80 mg + aliskiren 300 mg - (B) telmisartan 80 mg + eplerenon 50 mg - (C) telmisartan 160 mg
  Interventions: Drug: aliskiren, eplerenon, telmisartan
- B - A - C (Active Comparator): (A) telmisartan 80 mg + aliskiren 300 mg - (B) telmisartan 80 mg + eplerenon 50 mg - (C) telmisartan 160 mg
  Interventions: Drug: aliskiren, eplerenon, telmisartan
- A - B - C (Active Comparator): (A) telmisartan 80 mg + aliskiren 300 mg - (B) telmisartan 80 mg + eplerenon 50 mg - (C) telmisartan 160 mg
  Interventions: Drug: aliskiren, eplerenon, telmisartan

INTERVENTIONS:
Drug: aliskiren, eplerenon, telmisartan — aliskiren (Rasilez 300 mg, Novartis Europharm eplerenon (Inspra 50 mg, Pfizer Europe) telmisartan (Micardis 80 mg, Boehringer Ingelheim)

SUMMARY:
The main purpose of the study is to compare the effects of three different types of RAAS blockade on 24 hours proteinuria in patients with non-diabetic chronic kidney disease.

DETAILED DESCRIPTION:
Pharmacological blockade of the renin-angiotensin-aldosterone system (RAAS) is the main target of therapy to reduces both proteinuria and the rate of decline of the glomerular filtration rate in non-diabetic chronic renal diseases. Despite recent progress, however, there is still no optimal therapy that can stop the progression of these nephropathies. Therefore, it is necessary to optimize such treatment for further improving renal outcome.

The aim of the present study was to compare the effects of three different types of RAAS blockade: (1) mineralocorticoid receptor blocker (MRB) + angiotensin receptor antagonist (ARA); (2) direct renin inhibitor (DRI) + ARA and (3) double maximal dose of ARA on 24 hours proteinuria in patients with non-diabetic chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* chronic non-diabetic proteinuric nephropathy
* chronic kidney disease stage 1-3
* stable proteinuria above 500 mg/24 hours
* blood pressure above 125/75 mmHg and below 150/95 mmHg
* no steroids or other immunosuppressive treatment for a minimum of six months before the study

Exclusion Criteria:

* unstable coronary heart disease
* decompensated congestive heart failure in the previous 6 months
* episode of malignant hypertension or stroke in the history
* diabetes
* creatinine clearance below 30 ml/min
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference in urinary albumin-to-creatinine ratio (UACR) between treatment arms | baseline and the end of 8 week treatments
  changes of UACR

SECONDARY OUTCOMES:
Difference in transforming growth factor beta (TGF-beta) between treatment arms | baseline and the end of 8 week treatments
  Changes of urinary excretion of transforming growth factor beta (TGF-beta)
Difference in serum potassium and creatinine between treatment arms | baseline and the end of 8 week treatments

CONTACTS AND LOCATIONS:
Overall Officials: Bolesław Rutkowski, Professor, Principal Investigator — Departmen of Nephrology, Transplantation adn Internal Medicine, Medical University of Gdańsk, Poland